CLINICAL TRIAL: NCT03085238
Title: Safety and Performance of Metastatic Tumor Cell Trap Device in Patients With Advanced Ovarian Cancer
Brief Title: Metastatic Tumor Cell Trap Device in Patients With Advanced Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTrap, Inc. (Industry)
Collaborators: MedPass International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTRAP-2016-01
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Ovarian Cancer Stage IIIC; Ovarian Cancer Stage IV
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, non-blinded, single-arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- M-Trap (Experimental)
  Interventions: Device: M-Trap

INTERVENTIONS:
Device: M-Trap — Device(s) will be surgically implanted in the peritoneal cavity. Up to three (3) M-Trap devices will be surgically implanted via laparotomy in the right and left paracolic (pelvic) gutters and behind segment 6 of the liver within the peritoneal cavity of the patient at the time of surgical resection. Patients will receive standard platinum-based chemotherapy. If the cancer is diagnosed to have recurred, M-Trap devices with captured tumor cells will be removed via minimally invasive surgery (laparoscopy).

SUMMARY:
M-Trap is an implantable medical device designed to capture disseminated tumor cells (DTCs). It is intended for use in advanced-stage ovarian cancer patients. The study objective is to assess the safety and the performance of the M-Trap device.

ELIGIBILITY:
Inclusion Criteria:

1. Is a female ≥18 years old.
2. Presents with a diagnosis of Stage IIIC ovarian cancer.
3. Presents with high-grade serous carcinoma.
4. Has one of the following:

   1. Visible residual tumor ≤1 cm after primary tumor debulking surgery.
   2. Three cycles of neoadjuvant chemotherapy and complete resection after interval tumor debulking surgery.
   3. Three cycles of neoadjuvant chemotherapy and visible residual tumor ≤1 cm after interval tumor debulking surgery.
5. ECOG performance status of 0 or 1.
6. Is willing to comply with required follow-up study visits.
7. Is willing and able to provide written informed consent.

Exclusion Criteria:

1. Has a life expectancy of <3 months.
2. Is pregnant, as confirmed through a blood test prior to any study procedure, planning on becoming pregnant during the study, or is lactating.
3. Will be receiving intraperitoneal chemotherapy.
4. Has undergone prior treatment with abdominal and/or pelvic radiotherapy.
5. Has significant active concurrent medical illnesses including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Presence of central nervous system or cerebral metastases.
7. Recurrent ovarian cancer.
8. Complete resection with no residual tumor after primary tumor debulking surgery.
9. Suboptimal resection with >1 cm residual tumor after primary or interval tumor debulking surgery.
10. Is simultaneously enrolled in another investigational study.
11. Has a history of cancer within 5 years other than in-situ uterine cervix cancer or non-melanoma skin cancer.
12. Has a known hypersensitivity to carboplatin or paclitaxel.
13. Is concurrently using other antineoplastic agents.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gil-Moreno, MD, Principal Investigator — Hospital Vall d'Hebron
Locations (8):
- Spain (8):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Castellon University General Hospital, Castelló
  - MD Anderson Cancer Center, Madrid
  - Hospital La Paz Madrid, Madrid
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Valencia-Hospital General, Valencia
  - Hospital Universitrio y Politècnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective, multi-center, non-blinded, single-arm study
Groups:
- M-Trap: M-Trap: Device(s) will be surgically implanted in the peritoneal cavity.
Period: Overall Study
Arm/Group | M-Trap
Started | 23
1 Month | 23
3 Months | 22
6 Months | 19
9 Months | 16
12 Months | 14
15 Months | 11
18 Months | 7
Completed | 19
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | M-Trap
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 23
Ovarian Cancer Stage [Count of Participants; unit: Participants] — Staging is the process of finding out how much cancer is in a person's body and where it's located.
  Stage IIIC: Cancer has spread to the peritoneum and the cancer in the peritoneum is larger than 2 centimeters and/or cancer has spread to lymph nodes in the abdomen.
  Stage IVA: Cancer cells are found in extra fluid that has built up around the lungs.
  Stage IVB: Cancer has spread to organs and tissues outside the abdomen, including lymph nodes in the groin.
  Participants
    IIIC | 18
    IVA | 1
    IVB | 4
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group GRADE 0 Fully active, able to carry on all pre-disease performance without restriction GRADE 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature GRADE 2 Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours GRADE 3 Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours GRADE 4 Completely disabled; cannot carry on any selfcare; totally confined to bed or chair GRADE 5 Dead
  Participants
    Grade 0 | 16
    Grade 1 | 7
Pregnancy [Count of Participants; unit: Participants]
  Negative pregnancy test | 2
  Prior hysterectomy | 3
  Post-menopause | 18
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: 1 missing
  kg/m^2
    number analyzed (Participants) | 22
    (all) | 25.8 (3.7)
Type of debulking procedure [Count of Participants; unit: Participants] — Primary debulking has no chemotherapy treatment prior to the debulking surgery. Interval debulking has 3 to 4 rounds of chemotherapy treatment prior to the debulking surgery with the aim of reducing the tumor burden prior to surgery.
  Participants
    Primary | 8
    Interval with 3 rounds of chemotherapy | 11
    Interval with 4 rounds of chemotherapy | 4
Pre-debulking PCI [Mean (Standard Deviation); unit: scores on a scale] — Peritoneal cancer index (PCI) - assesses extent of peritoneal cancer in peritoneal cavity. Peritoneal cavity is divided in 13 well-defined regions. In each region, the size of the largest tumor nodule is measured. If no tumor is visualized, score is "0". If the largest tumor nodule is smaller than 0.5 cm, score is "1". If tumor measures between 0.5 cm and 5 cm, score is "2". If lesion is larger than 5 cm, the score is "3". If layering or a confluence of multiple small tumor nodules, score is "3". PCI is calculated by adding the scores of all regions together with a max of 39 (13×3). Population: Analysis on complete population and sub-analysis by type of debulking surgery.
  scores on a scale
    All patients | 17.8 (8.3)
    Primary debulking: number analyzed (Participants) | 8
    Primary debulking | 25.5 (3.4)
    Interval debulking: number analyzed (Participants) | 15
    Interval debulking | 13.7 (7.1)
Post-debulking PCI [Mean (Standard Deviation); unit: scores on a scale] — Peritoneal cancer index (PCI) - assesses extent of peritoneal cancer in peritoneal cavity. Peritoneal cavity is divided in 13 well-defined regions. In each region, the size of the largest tumor nodule is measured. If no tumor is visualized, score is "0". If the largest tumor nodule is smaller than 0.5 cm, score is "1". If tumor measures between 0.5 cm and 5 cm, score is "2". If lesion is larger than 5 cm, the score is "3". If layering or a confluence of multiple small tumor nodules, score is "3". PCI is calculated by adding the scores of all regions together with a max of 39 (13×3). Population: Measure Analysis Population Description: Analysis on complete population and sub-analysis by type of debulking surgery.
  scores on a scale
    All patients | 1.3 (1.5)
    Primary debulking: number analyzed (Participants) | 8
    Primary debulking | 2.7 (1.1)
    Interval debulking: number analyzed (Participants) | 15
    Interval debulking | 0.6 (1.1)
Pre-operative serum albumin [Mean (Standard Deviation); unit: g/dl] — Population: Data not recorded for two patients.
  g/dl
    number analyzed (Participants) | 21
    (all) | 6.5 (8.9)
Pre-operative hemoglobin [Mean (Standard Deviation); unit: g/dl] | 11.3 (1.4)
Total number of extended procedures [Count of Participants; unit: Participants] — Total number of extended procedures per the Patankar definition. Extended procedures of interest included lymphadenectomy, small bowel resection, colectomy, rectosigmoid resection, hepatic resection, bladder resection, diaphragm resection and cytoreduction.
  Participants
    1 extended procedure | 1
    2 extended procedures | 8
    3 or more extended procedures | 14

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Participants With Freedom From Device and Procedure-related Major Adverse Events
Description: The primary objective is to demonstrate that the safety of M-Trap, as measured by freedom from device- and procedure-related major adverse events through 6-months post-implantation, is non-inferior to historical controls (Patankar 2015). Freedom from device and procedure-related major adverse events is defined as severe complications based on Clavian Class IV complications, through 6-months post-implantation, including shock, cardiac arrest, myocardial infarction, pulmonary embolism, prolonged intubation, unplanned reintubation, or adverse events leading to removal of the device, including infection, seroma formation, mesh migration, bowel obstruction, adhesions, and local cancer progression through the abdominal wall at M-Trap suture sites.
Time Frame: 6 months
Population: All enrolled patients
Measure: Count of Participants; unit: Participants
Groups:
- M-Trap: M-Trap: Device(s) will be surgically implanted in the peritoneal cavity at time of surgical debulking.
Arm/Group | M-Trap
Number analyzed (Participants) | 23
Participants | 18
Statistical Analysis 1: Comparison: M-Trap; H0: M-Trap freedom MAE incidence <= 90% - Non-inferiority margin (25%); Test type: Non-Inferiority — The primary safety endpoint will be analyzed using a unilateral one sample test for binomial proportion at the 5% level; p = 0.1309, unilateral one sample test for binomial

2. Primary Outcome: Safety: Number of Participants With Freedom From Device and Procedure-related Major Adverse Events
Description: An additional analysis was performed to assess safety of M-Trap in comparison to historical controls at a comparable 30 day timepoint, as measured by freedom from device- and procedure-related major adverse events through 30 days post-implantation. Freedom from device and procedure-related major adverse events is defined as severe complications based on Clavian Class IV complications, through 30-days post-implantation, including shock, cardiac arrest, myocardial infarction, pulmonary embolism, prolonged intubation, unplanned reintubation, or adverse events leading to removal of the device, including infection, seroma formation, mesh migration, bowel obstruction, adhesions, and local cancer progression through the abdominal wall at M-Trap suture sites, adjusted based on the breakdown of the historical control population by number of extended procedures
Time Frame: 30 days
Population: All enrolled patients
Measure: Count of Participants; unit: Participants
Arm/Group | M-Trap
Number analyzed (Participants) | 23
Participants | 20
Statistical Analysis 1: Comparison: M-Trap; H0: M-Trap freedom MAE incidence <= 90% - Non-inferiority margin (25%); Test type: Non-Inferiority — The primary safety endpoint will be analyzed using a unilateral one sample test for binomial proportion at the 5% level; p = .0181, unilateral one sample test for binomial

3. Primary Outcome: Performance: Number of Participants With Histological Evidence of Tumor Cell Capture
Description: Histological evidence of tumor cell capture in at least one device in patients who underwent successful device removal
Time Frame: Time of device removal, an average of 13.3 months
Population: Assessment was completed in all patients who underwent successful device removal.
Measure: Count of Participants; unit: Participants
Groups:
- Platinum Resistant, Recurrent Patients: Tumor cell capture in at least one device in patients determined to be recurrent and platinum-resistant
- Platinum Sensitive, Recurrent Patients: Tumor cell capture in at least one device in patients determined to be recurrent and platinum-sensitive
- Non-recurrent: Tumor cell capture in at least one device in patients who did not demonstrate recurrence
- All Recurrent Patients: Tumor cell capture in at least one device in patients determined to be recurrent
- All Patients: Tumor cell capture in at least one device in all patients
Arm/Group | Platinum Resistant, Recurrent Patients | Platinum Sensitive, Recurrent Patients | Non-recurrent | All Recurrent Patients | All Patients
Number analyzed (Participants) | 4 | 9 | 8 | 13 | 21
Participants | 2 | 6 | 2 | 8 | 10

4. Secondary Outcome: Safety: Number of Participants With Device-related Long-term Adverse Event Reporting
Description: Device-related long-term adverse events and serious adverse events reported through 18 months
Time Frame: 18 months
Population: All enrolled patients
Measure: Count of Participants; unit: Participants
Arm/Group | M-Trap
Number analyzed (Participants) | 23
Participants | 1

5. Secondary Outcome: Safety: Number of Participants With Procedure-related Long-term Adverse Event Reporting
Description: Procedure-related long-term adverse events and serious adverse events reported through 18 months
Time Frame: 18 months
Population: All enrolled patients
Measure: Count of Participants; unit: Participants
Arm/Group | M-Trap
Number analyzed (Participants) | 23
Participants | 21

6. Secondary Outcome: Performance: Disease Focalization Score Categorized as I, I or II, I or II or III, and I or II or III or IV by Recurrence Status
Description: Disease focalization score - Disease focalization scores of I, II, III, IV, or V were assigned by the evaluating clinician, representing the approximate percentage 100%, 75%, 50%, 25%, or 0%, respectively, of recurrent tumor contained in the M-Trap device. Results are presented as described in secondary objective: patient count of score I; score I or II; score I, II or III; score I, II, III or IV; or No focalization.
Time Frame: Time of recurrence, an average of 14.5 months
Population: All patients with disease focalization scores reported
Measure: Count of Participants; unit: Participants
Groups:
- M-Trap Platinum Resistant Recurrent: Tumor cell capture in at least one device in patients determined to be recurrent and platinum-resistant
- Non-recurrent: Tumor cell capture in at least one device in patients determined to be non-recurrent
- All Recurrent Patients: Tumor cell capture in at least one device in all patients determined to be recurrent
Arm/Group | M-Trap Platinum Resistant Recurrent | Platinum Sensitive, Recurrent Patients | Non-recurrent | All Recurrent Patients | All Patients
Number analyzed (Participants) | 4 | 10 | 7 | 14 | 21
Participants
  I | 0 | 0 | 0 | 0 | 0
  I or II | 0 | 0 | 0 | 0 | 0
  I, II or III | 0 | 1 | 0 | 1 | 1
  I, II, III or IV | 2 | 7 | 0 | 9 | 9
  No focalization | 2 | 2 | 7 | 4 | 11

7. Other Pre Specified Outcome: Number of Devices Implanted
Description: Number of devices implanted at conclusion of debulking surgery.
Time Frame: Immediately post-procedure
Population: All patients
Measure: Count of Participants; unit: Participants
Arm/Group | M-Trap
Number analyzed (Participants) | 23
Participants
  2 devices | 1
  3 devices | 22

8. Other Pre Specified Outcome: Disease Focalization Score by Recurrence Status
Description: Disease focalization score - Disease focalization scores of I, II, III, IV, or V were assigned by the evaluating clinician, representing the approximate percentage 100%, 75%, 50%, 25%, or 0%, respectively, of recurrent tumor contained in the M-Trap device
Time Frame: Time of recurrence, an average of 14.5 months
Population: All patients with disease focalization scores reported
Measure: Count of Participants; unit: Participants
Arm/Group | M-Trap Platinum Resistant Recurrent | Platinum Sensitive, Recurrent Patients | Non-recurrent | All Recurrent Patients | All Patients
Number analyzed (Participants) | 4 | 10 | 7 | 14 | 21
Participants
  I (100% focalized) | 0 | 0 | 0 | 0 | 0
  II (~75% focalized | 0 | 0 | 0 | 0 | 0
  III (~50% focalized) | 0 | 1 | 0 | 1 | 1
  IV (~25% focalized) | 2 | 6 | 0 | 8 | 8
  V (no focalization) | 2 | 3 | 7 | 5 | 12

9. Other Pre Specified Outcome: Number of Participants With Reasons for Device Removal
Description: Reason that device removal was planned, regardless of whether or not it was completed.
Time Frame: Time of device removal, an average of 13.3 months
Population: All enrolled patients
Measure: Count of Participants; unit: Participants
Groups:
- M-Trap: M-Trap: Device(s) will be surgically implanted in the peritoneal cavity at the time of surgical debulking.
Arm/Group | M-Trap
Number analyzed (Participants) | 23
Participants
  Device-related adverse event necessitating removal | 1
  Disease progression | 15
  Final 18-month post-implantation time point | 5
  Major adverse event not related with the device | 1
  Death prior to removal | 1

10. Post Hoc Outcome: Tumor Cell Infiltration
Description: Estimate of tumor cell infiltration into the device based on histopathological analysis of devices from recurrent patients who underwent successful device removal. Percentage of device was determined by analysis of one slide from one tissue block (0.3 cm thick), by considering the amount of tumor cells in comparison to the total number of cells present in the slide when analyzed using image analysis with a digital slide scanner [Membrane Quant Module, Panoramic 250 FLASH II 2.0 (3D HISTEC)].
Time Frame: Time of recurrence, an average of 14.5 months
Population: Recurrent patients who underwent successful device removal
Measure: Mean (Standard Deviation); unit: percentage of device
Arm/Group | M-Trap
Number analyzed (Participants) | 13
percentage of device | 1.7 (2.5)

ADVERSE EVENTS:
Time Frame: 18 months
Description: Any adverse event (AE) observed was fully investigated by the Investigator and classified in line with the definitions of the ISO 14155:2011. AEs were collected from patients and their medical records at each follow-up interval (discharge, 1 month, 3 months, 6 months, 9 months, 12 months, 15 months, and 18 months).
Arm/Group | M-Trap
All-Cause Mortality (participants affected / at risk) | 2/23
Serious Adverse Events (participants affected / at risk) | 11/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M-Trap (N=23)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Procedural hemorrhage; disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1)
Intestinal anastomosis complication (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (3)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Pancreatic fistula (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Escherichia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3)
Post-operative fever (Injury, poisoning and procedural complications) | 1 (1)
Post-operative respiratory failure (Injury, poisoning and procedural complications) | 1 (2)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1)
Staphylococcal bacteraemia; Intervertebral discitis (Injury, poisoning and procedural complications) | 1 (1)
Bronchoplegia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Distributive shock (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M-Trap (N=23)
Abdominal pain (Gastrointestinal disorders) | 9 (12)
Vomiting (Gastrointestinal disorders) | 4 (4)
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Procedural hemorrhage (Injury, poisoning and procedural complications) | 13 (13)
Neurotoxicity (Injury, poisoning and procedural complications) | 4 (6)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Postoperative renal failure (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4)
Diarrhoea infectious (Infections and infestations) | 2 (2)
Bronchitis (Infections and infestations) | 1 (2)
Abdominal abscess (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Pyelonephritis fungal (Infections and infestations) | 1 (1)
Subdiaphragmatic abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (5)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Asthenia (General disorders) | 4 (4)
Chest pain (General disorders) | 1 (1)
Condition aggravated (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Febrile neutropenia (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Edema (General disorders) | 1 (1)
Edema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Onycholysis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Breast discharge (Reproductive system and breast disorders) | 1 (2)
Ovarian vein thrombosis (Reproductive system and breast disorders) | 1 (1)
Vaginal fistula (Reproductive system and breast disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Anemia; transfusion (Blood and lymphatic system disorders) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1)
Goitre (Endocrine disorders) | 1 (1)
Vomiting; diarrhea (Gastrointestinal disorders) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Lymphocele (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT03085238/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/38/NCT03085238/SAP_001.pdf